CLINICAL TRIAL: NCT04997161
Title: An Open-Label, Randomised, Controlled, Parallel-Design, Multicentre, Phase IV Study of Sodium Zirconium Cyclosilicate and Enhanced Nutrition Advice Compared to Standard of Care in Dialysis Patients With Hyperkalaemia (GRAZE)
Brief Title: Study of SZC and Enhanced Nutrition Advice Compared to SoC in Dialysis Patients With Hyperkalaemia
Acronym: GRAZE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: There is disconnect between dietary guidelines to limit potassium intake in dialysis and clinical practice. The number of unknowns and differences make the results unlikely to be translatable into clinical practice and will not benefit patients.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9480C00014; 2021-000457-81 (EudraCT Number)
Record Dates: First submitted 2021-06-16; First posted 2021-08-09 (Actual); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Hyperkalaemia
Keywords: Hyperkalaemia; Dialysis Patients
MeSH Terms: conditions — Hyperkalemia | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Intervention Model Description: Parallel: Participants are assigned to two groups in parallel for the duration of the study.
  Following 7-day screening, all participants who are enrolled will begin an up to 1-month HK Treatment Phase with SZC as per local label. Participants will receive dietary advice consistent with SoC at that site, including K+ restriction. A 4-month Diet Comparison Phase will begin next with participants being randomised to either continue taking SZC, which can be titrated as needed to maintain target S-K+ , and receive enhanced nutritional advice to consume fruit and vegetables (SZC arm), or SZC will be withdrawn and participants will receive SoC, including dietary K+ restriction (SoC arm).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SZC arm with enhanced dietary advice (Experimental): Participants will continue taking Sodium Zirconium Cyclosilicate (SZC), which can be titrated up or down to maintain S-K+ in the range 3.5-5.5 mmol/L; participants will also receive enhanced nutritional advice to consume fruit and vegetables. Advice will be provided by dietitians at study visits and by Noom app between visits.
  Interventions: Drug: Sodium Zirconium Cyclosilicate (SZC); Other: Enhanced dietary advice
- SoC arm with standard dietary advice (Other): SZC will be withdrawn and participants will receive SoC as per site practice, including dietary K+ restriction. Dietary advice will be given by dietitians at study visits and by Noom app between study visits.
  Interventions: Other: Standard dietary advice including K+ restriction.

INTERVENTIONS:
Drug: Sodium Zirconium Cyclosilicate (SZC) — Participants in the active arm will receive SZC dosed as per the local label to control hyperkalaemia and maintain normokalaemia.
  Other Names: SZC
  Arms: SZC arm with enhanced dietary advice
Other: Enhanced dietary advice — Participants will receive enhanced dietary advice in addition to taking SZC. This will include advice from dietitians to consume fruit and vegetables. Participants will be encouraged to consume up to 70 mmol K+ per day.
  Arms: SZC arm with enhanced dietary advice
Other: Standard dietary advice including K+ restriction. — Participants randomised to the SoC arm of the Diet Comparison Phase will receive standard dietary advice including K+ restriction.
  Other Names: Standard dietary advice
  Arms: SoC arm with standard dietary advice

SUMMARY:
Prescribing Sodium zirconium cyclosilicate (SZC) with enhanced nutritional advice to participants with hyperkalaemia on haemodialysis will reduce serum K+ (S-K+ ) and enable the consumption of more fruit and vegetables and more satisfying diet. The study aims to show that participants using SZC achieve S-K+ reduction as well as participants on SoC (other than K+ binders), without the need for restricting K+ in the diet.

DETAILED DESCRIPTION:
This is a Phase IV, randomised, controlled, open-label, parallel-group, multicentre, prospective study to evaluate the effect of the combination of SZC and enhanced nutritional advice to consume fruit and vegetables as compared to SoC in reducing S-K+ levels in participants with hyperkalaemia on haemodialysis. Following 7-day screening, all participants who are enrolled will begin an up to 1-month HK Treatment Phase with SZC as per local label. Participants will receive dietary advice consistent with SoC at that site, including K+ restriction. A 4-month Diet Comparison Phase will begin next with participants being randomised to either continue taking SZC, which can be titrated as needed to maintain target S-K+ , and receive enhanced nutritional advice to consume fruit and vegetables (SZC arm), or SZC will be withdrawn and participants will receive SoC, including dietary K+ restriction (SoC arm).

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥18 years of age at the time of signing the informed consent.
2. Participants with prevalent HK (S-K+ >5.5 mmol/L at the end of LIDI) not requiring acute treatment.
3. Receiving haemodialysis 3 times a week with stable vascular access for at least 3 months before screening visit.
4. Participants who have and are able and willing to use smart phone (android or iOS) nutrition app.
5. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   * Female participants of childbearing potential must have a negative pregnancy test.
   * Female participants must be 1 year post-menopausal, surgically sterile, or using 1 highly effective form of birth control (defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly). They should have been stable on their chosen method of birth control for a minimum of 3 months before entering the study and willing to remain on the birth control until 12 weeks after the last dose.
6. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and in the protocol.

Exclusion Criteria:

1. As judged by the investigator or sponsor, any medical condition (including active, clinically significant infection) that may pose a safety risk to the participant in this study, may confound safety or efficacy assessments and jeopardise the quality of data, or may interfere with study participation.
2. Myocardial infarction, acute coronary syndrome (ST-elevation myocardial infarction, non-ST-elevation myocardial infarction, or unstable angina), stroke, seizure, thrombotic/thromboembolic event (eg, deep vein thrombosis or pulmonary embolism, but excluding vascular access thrombosis), percutaneous transluminal coronary angioplasty, or coronary artery bypass graft within 12 weeks prior to screening visit.
3. Severe leucocytosis (>20 × 109 /L) or thrombocytosis (≥450 × 109 /L) during screening.
4. Polycythaemia (haemoglobin >14 g/dL) during screening.
5. Severe constipation, bowel obstruction, post-operative motility disorders.
6. Scheduled date for living donor kidney transplant.
7. Participants with a life expectancy of less than 6 months.
8. Females of childbearing potential, unless using contraception as detailed in the protocol or sexually abstinent.
9. Currently pregnant (confirmed with positive pregnancy test) or breast-feeding.
10. Presence of cardiac arrhythmias or conduction defects that require immediate treatment at HCP discretion.
11. History of alcohol or drug abuse within 2 years prior to screening visit.
12. History of QT prolongation associated with other medications that required discontinuation of that medication.
13. Congenital long QT syndrome or QT interval corrected for heart rate (QTc) using Fridericia's method (QTcF) >550 ms.
14. Symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Subjects with atrial fibrillation controlled by medication are permitted.
15. If the participant has evidence of Coronavirus disease 2019 (COVID-19) within 2 weeks prior to screening (see Appendix D), the participant cannot be enrolled in the study.
16. Participants treated with SZC, sodium polystyrene sulfonate (SPS: Kayexalate™; Resonium™ A), calcium polystyrene sulfonate (CPS: Calcium Resonium™), or patiromer (Veltassa™) 1 within 4 weeks before screening.
17. Participants with a known hypersensitivity or previous anaphylaxis to SZC or any of the excipients of the product.
18. Participants unable to take oral SZC. Prior/Concurrent Clinical Study Experience
19. Participation in another clinical study with an investigational product administered during the month before screening2 .
20. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
21. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
22. Previous enrolment in the present study.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wittbrodt, PharmD, MPH, Study Director — AstraZeneca, Biopharmaceuticals Medical
Locations (1):
- Research Site, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Clinical Study Protocol-redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00014&attachmentIdentifier=26c9fb48-f14a-43a0-a51b-53e7c34bf64c&fileName=Clinical_Study_Protocol-redacted.pdf&versionIdentifier=
- See also: Statistical Analysis Plan-redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00014&attachmentIdentifier=224e8afa-bd15-4a63-a6fc-4368fd5e111d&fileName=Statistical_Analysis_Plan-redacted.pdf&versionIdentifier=
- See also: CSR synopsis-redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00014&attachmentIdentifier=71d57d2b-b5ef-4373-9ae4-d80f335467b2&fileName=CSR_synopsis-redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was randomised prior to study termination by sponsor
Groups:
- Overall Study: All enrolled participants
Period: Overall Study
Arm/Group | Overall Study
Started | 3
Randomized (Randomized to receive SZC 5 g once daily orally until the end of Month 2 in addition to enhanced nutritional advice to consume fruit and vegetables.) | 1
Completed | 0
Not Completed | 3
Not completed — Study terminated by sponsor | 3

BASELINE CHARACTERISTICS:
Population: The baseline population includes the one participant randomized in this study.
Groups:
- Randomized Participants: All randomized participants
Arm/Group | Randomized Participants
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants] — Population: test
  Participants
    <=18 years | NA — As only one participant was randomized, baseline data is not presented in order to protect participant confidentiality.
    Between 18 and 65 years | NA — As only one participant was randomized, baseline data is not presented in order to protect participant confidentiality.
    >=65 years | NA — As only one participant was randomized, baseline data is not presented in order to protect participant confidentiality.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — As only one participant was randomized, baseline data is not presented in order to protect participant confidentiality.
  Male | NA — As only one participant was randomized, baseline data is not presented in order to protect participant confidentiality.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — As only one participant was randomized, baseline data is not presented in order to protect participant confidentiality.
  Asian | NA — As only one participant was randomized, baseline data is not presented in order to protect participant confidentiality.
  Native Hawaiian or Other Pacific Islander | NA — As only one participant was randomized, baseline data is not presented in order to protect participant confidentiality.
  Black or African American | NA — As only one participant was randomized, baseline data is not presented in order to protect participant confidentiality.
  White | NA — As only one participant was randomized, baseline data is not presented in order to protect participant confidentiality.
  More than one race | NA — As only one participant was randomized, baseline data is not presented in order to protect participant confidentiality.
  Unknown or Not Reported | NA — As only one participant was randomized, baseline data is not presented in order to protect participant confidentiality.

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Potassium
Description: Change in serum potassium taken at long interdialytic-dialysis interval visits Month 3, Month 4, and Month 5 compared to baseline
Time Frame: Baseline to Month 5
Population: Data were not collected as the study closed prior to the pre-specified Time Frame for analysis.
Arm/Group | Randomized Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Change From Baseline in Fruit and Vegetable Consumption Determined by Participant-reported Intake Using Noom App From Month 2 to Month 5
Description: Change from baseline in fruit and vegetable consumption determined by participant-reported intake using Noom app from Month 2 to Month 5
Time Frame: Month 2 to Month 5
Population: Data were not collected as the study closed prior to the pre-specified Time Frame for analysis.
Arm/Group | Randomized Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Effect of the Combination of Sodium Zirconium Cyclosilicate and Enhanced Nutritional Advice as Compared to Standard of Care on Participant-reported Chronic Kidney Disease Symptoms, Physical and Mental Health, and Satisfaction With Treatment
Description: Electronic versions of the following:
  Kidney Disease and Quality of Life-36 item (KDQOL-36; symptoms/problems, Physical Component Summary and Mental Component Summary, Burden of Kidney Disease and Effects of Kidney Disease)
  EuroQol-5 Dimensions-5 Levels (EQ-5D-5L)
  Abbreviated Treatment Satisfaction Questionnaire for Medication (9 items) (TSQM-9)
  Patients' Global Impression of Change (PGIC)
Time Frame: From study start to study end
Population: Data were not collected due to study early termination.
Arm/Group | Randomized Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: Effect of the Combination of Sodium Zirconium Cyclosilicate and Enhanced Nutritional Advice to Consume Fruit and Vegetables as Compared to Standard of Care in Maintaining Serum Potassium Levels
Description: Effect of the combination of sodium zirconium cyclosilicate and enhanced nutritional advice to consume fruit and vegetables as compared to standard of care in maintaining serum potassium levels within a range of 3.5 to 5.5 mmol/L, without requiring rescue therapy for hyperkalaemia.
  Binary response (responder/non-responder) with criteria that at least 66% of serum potassium values taken at long interdialytic-dialysis interval visits in Months 3, 4, and 5 fall between 3.5 and 5.5 mmol/L.
  Receiving rescue therapy or a potassium binder for hyperkalaemia during the final 3 months of the study was to result in a non-response.
Time Frame: From study start to study end
Population: Data were not collected as the study closed prior to the pre-specified Time Frame for analysis.
Arm/Group | Randomized Participants
Number analyzed (Participants) | 0

5. Secondary Outcome: Safety and Tolerability of Sodium Zirconium Cyclosilicate and Enhanced Nutritional Advice as Compared to Standard of Care
Description: Safety and tolerability were to be evaluated in terms of adverse events (AEs), vital signs, clinical laboratory, interdialytic weight gain, and electrocardiograms.
  Assessments related to AEs covered occurrence/frequency, relationship to sodium zirconium cyclosilicate as assessed by Investigator, intensity, seriousness, death, and AEs leading to discontinuation of sodium zirconium cyclosilicate.
Time Frame: From study start to study end
Population: Data were not collected due to study early termination.
Arm/Group | Randomized Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Assessed for a total of up to 179 days from screening/enrollment visit (Visit 1).
Arm/Group | Randomized Participants
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The study was terminated by the sponsor with only 1 participant randomized. There was disconnect between dietary guidelines to limit potassium intake in dialysis and clinical practice.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall be entitled to publish the results of, or make presentations related to, the Study, provided that any publications or presentations to be made within 2 years of completion of the Study shall require the Sponsor's prior written consent.

The Investigator will provide the Sponsor with copies of any materials relating to the study or developed technologies that they intend to publish or present at least 30 days in advance of publication, submission, or presentation.

DOCUMENTS (2):
  • Study Protocol (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT04997161/Prot_002.pdf
  • Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT04997161/SAP_001.pdf